CLINICAL TRIAL: NCT02323334
Title: Single- and Multiple-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY3202626
Brief Title: A Study of LY3202626 in Healthy Participants and Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 15562; I7X-EW-LLCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-12-08; First posted 2014-12-23 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — LY3202626; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (17):
- Part A Cohort 1 Sequence1: 0.1mg, 1.6mg, Placcebo; 15mg (Placebo Comparator): Part A Cohort 1 involved healthy participants and was comprised of 4 treatment periods with a washout period of approximately 14 days between doses.
  Period 1: 0.1mg LY3202626 Period 2: 1.6mg LY3202626 Period 3: 15 mg placebo (PBO) Period 4: 15mg LY3202626.
  Interventions: Drug: LY3202626; Drug: Placebo (Part A, B, C)
- Part A Cohort 1 Sequence 2: 0.1mg, PBO, 15mg, 15mg (Experimental): Part A Cohort 1 involved healthy participants and comprised of 4 treatment periods with a washout period of approximately 14 days between doses.
  Period 1: 0.1mg Period 2: PBO Period 3: 15mg LY3202626 Period 4: 15mg LY3202626.
  Interventions: Drug: LY3202626; Drug: Placebo (Part A, B, C)
- Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, Placebo (Experimental): Part A Cohort 1 involved healthy participants and comprised of 4 treatment periods with a washout period of approximately 14 days between doses.
  Period 1: PBO Period 2: 1.6mg LY3202626 Period 3: 15mg LY3202626 Period 4: PBO.
  Interventions: Drug: LY3202626; Drug: Placebo (Part A, B, C)
- Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO, 0.4mg/Itraconazole (Experimental): Part A Cohort 2 involved healthy participants and comprised of 4 treatment periods with a washout period of approximately 14 days between doses.
  Period 1: 0.4mg LY3202626 Period 2: 5mg LY3202626 Period 3: 45mg, PBO Period 4: 0.4mg LY3202626/200mg Itraconazole.
  Interventions: Drug: LY3202626; Drug: Placebo (Part A, B, C)
- Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/Itra (Experimental): Part A Cohort 2 involved healthy participants and comprised of 4 treatment periods with a washout period of approximately 14 days between doses.
  Period 1: 0.4mg LY3202626 Period 2: 5mg, PBO Period 3: 45mg LY3202626 Period 4: 0.4mg LY3202626/200mg Itraconazole.
  Interventions: Drug: LY3202626; Drug: Placebo (Part A, B, C); Drug: Itraconazole
- Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra (Experimental): Part A Cohort 2 involved healthy participants and was comprised of 4 treatment periods with a washout period of approximately 14 days between doses.
  Period 1: 0.4mg, PBO Period 2: 5mg LY3202626 Period 3: 45mg LY3202626 Period 4: 0.4mg LY3202626/200mg Itraconazole.
  Interventions: Drug: LY3202626; Drug: Placebo (Part A, B, C); Drug: Itraconazole
- Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted (Experimental): Part A Cohort 3 involved healthy participants and was comprised of two treatment periods with a washout period of approximately 14 days between doses. Single dose of 10mg LY3202626 given PO in Period 1 and 2. Period 1: Fed 2: Fasted.
  Interventions: Drug: LY3202626
- Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed (Experimental): Part A Cohort 3 involved healthy participants and was comprised of two treatment periods with a washout period of approximately 14 days between doses. Single dose 10mg LY3202626 given PO in Period 1 and 2. Period 1: Fasted 2: Fed.
  Interventions: Drug: LY3202626
- Part B Cohort 4: 1.6mg (Experimental): Part B Cohort 4 involved healthy participants and was comprised of one period. Single dose of 1.6mg LY3202626 given PO in Period 1. Dose determined by Part A.
  Interventions: Drug: LY3202626
- Part B Cohort 5: 10mg (Experimental): Part B Cohort 5 involved healthy participants and was comprised of one period. Single dose of 10mg LY3202626 given PO in Period 1. Dose determined by Part A.
  Interventions: Drug: LY3202626
- Part B Cohort 6: 26mg (Experimental): Part B Cohort 6 involved healthy participants and was comprised of one period. Single dose of 26mg LY3202626 given PO in Period 1. Dose determined by Part A.
  Interventions: Drug: LY3202626
- Part B Cohort 4, 5, 6: Placebo Comparator (Placebo Comparator): Part B Cohort 4,5,6 involved healthy participants and was comprised of one period. Single dose of PBO given PO in Period 1.
  Interventions: Drug: Placebo (Part A, B, C)
- Part C Cohort 7: 1mg (Experimental): Part C Cohort 7 involved healthy participants and was comprised of one period. 1mg LY3202626 given PO once daily for 14 days. Dose determined by Part B.
  Interventions: Drug: LY3202626
- Part C Cohort 8: 6mg (Experimental): Part C Cohort 8 involved healthy participants and was comprised of one period. 6mg LY3202626 was given PO once daily for 14 days. Dose determined by Part B.
  Interventions: Drug: LY3202626
- Part C Cohort 9: 26mg (Experimental): Part C Cohort 9 included healthy participants and was comprised of one period. 26mg LY3202626 was given PO once daily for 14 days. Dose determined by Part B.
  Interventions: Drug: LY3202626
- Part C Cohort 7, 8 ,9: Placebo Comparator (Placebo Comparator): Part C Cohort 7,8,9 involved healthy participants and was comprised of one period. Placebo given PO once daily for 14 days.
  Interventions: Drug: Placebo (Part A, B, C)
- Part D Cohort 10: 6mg (Experimental): Part D Cohort 10 involved participants with Alzheimer's disease and was comprised of one period. 6mg LY3202626 was given PO once daily for 14 days. Dose determined by Part B.
  Interventions: Drug: LY3202626

INTERVENTIONS:
Drug: LY3202626 — administered orally
  Arms: Part A Cohort 1 Sequence 2: 0.1mg, PBO, 15mg, 15mg; Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, Placebo; Part A Cohort 1 Sequence1: 0.1mg, 1.6mg, Placcebo; 15mg; Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO, 0.4mg/Itraconazole; Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/Itra; Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra; Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted; Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed; Part B Cohort 4: 1.6mg; Part B Cohort 5: 10mg; Part B Cohort 6: 26mg; Part C Cohort 7: 1mg; Part C Cohort 8: 6mg; Part C Cohort 9: 26mg; Part D Cohort 10: 6mg
Drug: Placebo (Part A, B, C) — administered orally
  Arms: Part A Cohort 1 Sequence 2: 0.1mg, PBO, 15mg, 15mg; Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, Placebo; Part A Cohort 1 Sequence1: 0.1mg, 1.6mg, Placcebo; 15mg; Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO, 0.4mg/Itraconazole; Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/Itra; Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra; Part B Cohort 4, 5, 6: Placebo Comparator; Part C Cohort 7, 8 ,9: Placebo Comparator
Drug: Itraconazole — administered orally
  Arms: Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/Itra; Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra

SUMMARY:
This study involves single and multiple doses of LY3202626 and will evaluate the effects of LY3202626 on the body. There will be 4 parts to this study. In Parts A and B, single increasing doses of LY3202626 will be given in capsule form. Part A will also include itraconazole given orally as a solution. Part A will last approximately 8-12 weeks. Part B will last approximately 5-6 weeks. In Parts C and D, participants will be dosed multiple days with the study drug. Part C will last approximately 11-14 weeks. Part D will last approximately 11-14 weeks and participants must have Alzheimer's Disease. Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* For Parts A, B, and C, are overtly healthy males or females (nonchildbearing potential), as determined by medical history and physical examination
* Have a body mass index (BMI) of 18 to 32 kilograms per square meter (kg/m^2)
* For Part D, present with Mild Cognitive Impairment (MCI) due to Alzheimer's Disease (AD) or mild to moderate AD
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures and research unit policies

Exclusion Criteria:

* Taking over-the-counter or prescription medication with the exception of vitamins or minerals
* Smoke more than 10 cigarettes per day
* Are unwilling or unable to refrain from eating any food or drinking any beverage containing grapefruit or grapefruit juice for at least 2 weeks prior to first dose until completion of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Cohort 1 Sequence 1: 0.1mg, 1.6mg, Placebo (PBO); 15mg: Part A Cohort 1 involved healthy participants and was comprised of 4 treatment periods. There was a washout period of approximately 14 days between doses.
  Period 1: 0.1mg LY3202626 Period 2: 1.6mg LY3202626 Period 3: 15 mg PBO Period 4: 15mg LY3202626
- Part A Cohort 1 Sequence 2: 1.6mg, PBO,15mg, 15mg: Part A Cohort 1 involved healthy participants and was comprised of 4 treatment periods. There was a washout period of approximately 14 days between doses.
  Period 1: 1.6mg LY3202626 Period 2: PBO Period 3: 15mg LY3202626 Period 4: 15mg LY3202626
- Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, PBO: Part A Cohort 1 involved healthy participants and was comprised of 4 treatment periods. There was a washout period of approximately 14 days between doses.
  Period 1: PBO Period 2: 1.6mg LY3202626 Period 3: 15mg LY3202626 Period 4: PBO
- Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO; 0.4mg/200mg Itra: Part A Cohort 2 involved healthy participants and was comprised of 4 treatment periods. Period 4 includes 0.4mg LY3202626 and 200mg Itraconazole (Itra). There was a washout period of approximately 14 days between doses.
  Period 1: 0.4mg LY3202626 Period 2: 5mg LY3202626 Period 3: 45mg PBO Period 4: 0.4mg LY3202626/200mg Itraconazole
- Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/200mg Itra: Part A Cohort 2 involved healthy participants and was comprised of 4 treatment periods. Period 4 includes 0.4mg LY3202626 and 200mg Itraconazole.There was a washout period of approximately 14 days between doses.
  Period 1: 0.4mg LY3202626 Period 2: 5mg PBO Period 3: 45mg LY3202626 Period 4: 0.4mg LY3202626/200mg Itraconazole
- Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra: Part A Cohort 2 involved healthy participants and was comprised of 4 treatment periods. Period 4 includes 0.4mg LY3202626 and 200mg Itraconazole. There was a washout period of approximately 14 days between doses.
  Period 1: 0.4mg PBO Period 2: 5mg LY3202626 Period 3: 45mg LY3202626 Period 4: 0.4mg LY3202626/200mg Itraconazole
- Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted: Part A Cohort 3 involved healthy participants and was comprised of two treatment periods. Single dose of 10mg LY3202626 given PO in Period 1 and 2. There was a washout period of approximately 14 days between doses.
  Period 1: Fed Period 2: Fasted
- Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed: Part A Cohort 3 involved healthy participants and was comprised of two treatment periods. Single dose 10mg LY3202626 given PO in Period 1 and 2.
  There was a washout period of approximately 14 days between doses.
  Period 1: Fasted Period 2: Fed
- Part B Cohort 4, 5, 6: PBO Comparator: Part B Cohort 4,5,6 involved healthy participants and was comprised of one period. Single dose of PBO given PO in Period 1.
- Part C Cohort 7, 8 ,9: PBO Comparator: Part C Cohort 7, 8, 9 involved healthy participants and was comprised of one period. PBO given PO once daily for 14 days.
Period: Period 1
Arm/Group | Part A Cohort 1 Sequence 1: 0.1mg, 1.6mg, Placebo (PBO); 15mg | Part A Cohort 1 Sequence 2: 1.6mg, PBO,15mg, 15mg | Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, PBO | Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO; 0.4mg/200mg Itra | Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/200mg Itra | Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra | Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted | Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed | Part B Cohort 4: 1.6mg | Part B Cohort 5: 10mg | Part B Cohort 6: 26mg | Part B Cohort 4, 5, 6: PBO Comparator | Part C Cohort 7: 1mg | Part C Cohort 8: 6mg | Part C Cohort 9: 26mg | Part C Cohort 7, 8 ,9: PBO Comparator | Part D Cohort 10: 6mg
Started | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 5 | 7 | 5 | 3 | 9 | 9 | 9 | 9 | 2
Received at Least One Dose of Study Drug | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 5 | 7 | 5 | 3 | 9 | 9 | 9 | 9 | 2
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 5 | 7 | 5 | 3 | 9 | 9 | 9 | 9 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A Cohort 1 Sequence 1: 0.1mg, 1.6mg, Placebo (PBO); 15mg | Part A Cohort 1 Sequence 2: 1.6mg, PBO,15mg, 15mg | Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, PBO | Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO; 0.4mg/200mg Itra | Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/200mg Itra | Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra | Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted | Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed | Part B Cohort 4: 1.6mg | Part B Cohort 5: 10mg | Part B Cohort 6: 26mg | Part B Cohort 4, 5, 6: PBO Comparator | Part C Cohort 7: 1mg | Part C Cohort 8: 6mg | Part C Cohort 9: 26mg | Part C Cohort 7, 8 ,9: PBO Comparator | Part D Cohort 10: 6mg
Started | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 0 (Part B was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part B was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part B was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part B was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part C was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part C was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part C was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part C was a single period conducted in parallel to Part A and received last dose in Period 1.) | 0 (Part D was a single period conducted in parallel to Part A and received last dose in Period 1.)
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A Cohort 1 Sequence 1: 0.1mg, 1.6mg, Placebo (PBO); 15mg | Part A Cohort 1 Sequence 2: 1.6mg, PBO,15mg, 15mg | Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, PBO | Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO; 0.4mg/200mg Itra | Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/200mg Itra | Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra | Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted | Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed | Part B Cohort 4: 1.6mg | Part B Cohort 5: 10mg | Part B Cohort 6: 26mg | Part B Cohort 4, 5, 6: PBO Comparator | Part C Cohort 7: 1mg | Part C Cohort 8: 6mg | Part C Cohort 9: 26mg | Part C Cohort 7, 8 ,9: PBO Comparator | Part D Cohort 10: 6mg
Started | 4 | 4 | 4 | 4 | 4 | 4 | 0 (Part A Cohort 3 Food Effect participated in Period 1 and Period 2 only.) | 0 (Part A Cohort 3 Food Effect participated in Period 1 and Period 2 only.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 4 | 3 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Part A Cohort 1 Sequence 1: 0.1mg, 1.6mg, Placebo (PBO); 15mg | Part A Cohort 1 Sequence 2: 1.6mg, PBO,15mg, 15mg | Part A Cohort 1 Sequence 3: PBO, 1.6mg, 15mg, PBO | Part A Cohort 2 Sequence 1:0.4mg, 5mg, PBO; 0.4mg/200mg Itra | Part A Cohort 2 Sequence 2: 0.4mg, PBO, 45mg. 0.4mg/200mg Itra | Part A Cohort 2 Sequence 3:PBO, 5mg, 45mg,0.4mg/200mg Itra | Part A Cohort 3 Sequence 1: Food Effect Fed/Fasted | Part A Cohort 3 Sequence 2: Food Effect Fasted/Fed | Part B Cohort 4: 1.6mg | Part B Cohort 5: 10mg | Part B Cohort 6: 26mg | Part B Cohort 4, 5, 6: PBO Comparator | Part C Cohort 7: 1mg | Part C Cohort 8: 6mg | Part C Cohort 9: 26mg | Part C Cohort 7, 8 ,9: PBO Comparator | Part D Cohort 10: 6mg
Started | 3 | 4 | 3 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 4 | 3 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Received at least one dose of study drug.
Groups:
- Part A Cohort 1: Escalating single dose given orally (PO)per randomly assigned treatment sequence of 0.1mg, 1.6mg, 15mg LY3202626 or placebo.
- Part A Cohort 2: Escalating single dose given PO per randomly assigned treatment sequence of 0.4mg, 5mg, or 45mg LY3202626, placebo.
  Some participants may also receive multiple doses of 200 mg of Itraconazole PO in 1 period with 0.4mg of LY3202626.
- Part A Food Effect Cohort 3: Single dose of 10mg LY3202626 given PO in Period 1 and Period 2 only.
- Part B Cohort 4: Single oral dose of 1.6mg LY3202626 or placebo given PO in Period 1. Dose determined by Part A.
- Part B Cohort 5: Single oral dose of 10mg LY3202626 or placebo given PO in in Period 1. Dose determined by Part A.
- Part B Cohort 6: Single oral dose of 26mg LY3202626 or placebo given PO in Period 1. Dose determined by Part A.
- Part C Cohort 7: Multiple oral doses of 1mg LY3202626 given PO once daily for 14 days. Dose determined by Part B.
- Part C Cohort 8; Part D Cohort 10: Multiple oral doses of 6mg LY3202626 given PO once daily for 14 days. Dose determined by Part B.
- Part C Cohort 9: Multiple oral doses of 26mg LY3202626 given PO once daily for 14 days. Dose determined by Part B.
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1 | Part A Cohort 2 | Part A Food Effect Cohort 3 | Part B Cohort 4 | Part B Cohort 5 | Part B Cohort 6 | Part C Cohort 7 | Part C Cohort 8 | Part C Cohort 9 | Part D Cohort 10 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 6 | 8 | 6 | 12 | 12 | 12 | 2 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (8.1) | 36.9 (8.4) | 39.0 (13.6) | 36.5 (12.4) | 43.0 (11.3) | 35.2 (7.2) | 37.5 (10.5) | 40.4 (8.1) | 40.5 (10.5) | 68.0 (2.8) | 38.70 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 10
  Male | 11 | 11 | 8 | 6 | 8 | 6 | 12 | 11 | 11 | 0 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3 | 0 | 1 | 3 | 2 | 3 | 3 | 0 | 18
  Not Hispanic or Latino | 10 | 11 | 9 | 6 | 7 | 3 | 10 | 9 | 9 | 2 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 4 | 0 | 0 | 0 | 4 | 4 | 4 | 2 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 2 | 1 | 1 | 3 | 3 | 1 | 0 | 18
  White | 3 | 4 | 5 | 4 | 7 | 5 | 4 | 5 | 7 | 0 | 44
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 6 | 8 | 6 | 12 | 12 | 12 | 2 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other nonserious Adverse Events (AE's), and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline to Study Completion (up to 14 weeks)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A, B, and C Placebo (PBO): Single dose placebo given PO in Part A and B. Multiple doses of PBO given PO in Part C.
- Part A 0.1mg LY3202626: Single dose of 0.1mg LY3202626 given PO Period 1 Cohort 1.
- Part A 0.4mg LY3202626: Single dose of 0.4mg LY3202626 given PO in Period 1 Cohort 2.
- Part A 0.4mg LY3202626 + 200mg Itraconazole: Single dose of 0.4mg LY3202626 +200mg Itraconazole given PO in Period 4 Cohort 2.
- Part C 1mg LY3202626 QD: Multiple daily dose of 1mg LY3202626 given PO once daily for 14 days.
- Part A and B 1.6mg LY3202626: Single dose of 1.6mg LY3202626 given PO in Period 2 Cohort 1 in Part A and Period 1 Part B.
- Part A 5mg LY3202626: Single dose of 5mg LY3202626 given PO in in Period 2 Cohort 2.
- Part C and D 6mg LY3202626 QD: Multiple daily dose of 6mg LY3202626 given PO once daily for 14 days.
- Part A, B and C 10mg LY3202626: Single dose of 10mg LY3202626 given PO in Part A and B. Multiple dose of 10mg LY3202626 given PO in Part C once daily for 14 days.
- Part A 15mg LY3202626: Single dose of 15mg LY3202626 given PO in Period 3 Cohort 1.
- Part B and C 26mg LY3202626: Single dose of 26mg LY3202626 given PO in Period 1 in Part B. Multiple daily dose of 26mg LY3202626 given PO once daily for 14 days in Part C.
- Part A 45mg LY3202626: Single dose of 45mg LY3202626 given PO in in Period 3 Cohort 2.
Arm/Group | Part A, B, and C Placebo (PBO) | Part A 0.1mg LY3202626 | Part A 0.4mg LY3202626 | Part A 0.4mg LY3202626 + 200mg Itraconazole | Part C 1mg LY3202626 QD | Part A and B 1.6mg LY3202626 | Part A 5mg LY3202626 | Part C and D 6mg LY3202626 QD | Part A, B and C 10mg LY3202626 | Part A 15mg LY3202626 | Part B and C 26mg LY3202626 | Part A 45mg LY3202626
Number analyzed (Participants) | 36 | 8 | 8 | 12 | 9 | 13 | 8 | 11 | 19 | 11 | 14 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY3202626
Description: Summary of PK parameters of LY3202626 in plasma following oral administration of single doses for Parts A and B and multiple doses for Part C.
Time Frame: Part A and B Day 1:Predose, 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours postdose; Part C Day 1:Predose, 0.5,1, 2, 4, 6, 8, and 12 hours postdose; Part C Day 14:Predose, 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, and 216 hours postdose
Population: All participants in Part A, B, and C who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A 0.1mg LY3202626: Single dose of 0.1mg LY3202626 given PO in Period 1 Cohort 1.
- Part A 1.6mg LY3202626: Single dose of 1.6mg LY3202626 given PO in Period 2 Cohort 1.
- Part A 5mg LY3202626: Single dose of 5mg LY3202626 given PO in Period 2 Cohort 2.
- Part A 45mg LY3202626: Single dose of 45mg LY3202626 given PO in Period 3 Cohort 2.
- Part B 1.6mg LY3202626: Single dose of 1.6mg LY3202626 given PO Period 1.
- Part B 10mg LY3202626: Single dose of 10mg LY3202626 given PO in Period 1.
- Part B 26mg LY3202626: Single dose of 26mg LY3202626 given PO in Period1.
- Part C 1mg LY3202626 QD: Multiple doses of 1mg LY3202626 given PO once daily for 14 days.
- Part C 6mg LY3202626 QD: Multiple doses of 6mg LY3202626 given PO once daily for 14 days.
- Part C 26mg LY3202626 QD: Multiple doses of 26mg LY3202626 given PO once daily for 14 days.
Arm/Group | Part A 0.1mg LY3202626 | Part A 0.4mg LY3202626 | Part A 1.6mg LY3202626 | Part A 5mg LY3202626 | Part A 15mg LY3202626 | Part A 45mg LY3202626 | Part B 1.6mg LY3202626 | Part B 10mg LY3202626 | Part B 26mg LY3202626 | Part C 1mg LY3202626 QD | Part C 6mg LY3202626 QD | Part C 26mg LY3202626 QD
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 8 | 5 | 7 | 5 | 8 | 9 | 9
nanograms per milliliter (ng/mL) | 0.169 (50) | 0.486 (81) | 2.89 (70) | 7.91 (56) | 21.3 (77) | 92.5 (47) | 2.90 (86) | 3.75 (176) | 36.1 (126) | 2.57 (2.5) | 11.2 (71) | 72.8 (61)

3. Secondary Outcome: PK: Area Under the Concentration Time Curve (AUC) of LY3202626
Description: Pharmacokinetic parameters for Part A and B were assessed on Day 1 using AUC 0-infinity (AUC0-inf). Pharmacokinetic parameters for Part C were assessed on Day 1 using AUC zero to time to last (AUC0-tlast), Day 14 using AUC steady state.
Time Frame: Part A and B Day 1: Predose, 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours postdose; Part C Day 1:Presdose, 0.5,1, 2, 4, 6, 8,12 hours postdose; Day 14: Predose, 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, and 216 hours postdose
Population: All participants in Parts A, B, and C who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram x hour/milliliter (ng*hr/mL)
Groups:
- Part B 1.6mg LY3202626: Single dose of 1.6mg LY3202626 given PO in Period 1.
- Part B 26mg LY3202626: Single dose of 26mg LY3202626 given PO in Period 1.
Arm/Group | Part A 0.1mg LY3202626 | Part A 0.4mg LY3202626 | Part A 1.6mg LY3202626 | Part A 5mg LY3202626 | Part A 15mg LY3202626 | Part A 45mg LY3202626 | Part B 1.6mg LY3202626 | Part B 10mg LY3202626 | Part B 26mg LY3202626 | Part C 1mg LY3202626 QD | Part C 6mg LY3202626 QD | Part C 26mg LY3202626 QD
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 8 | 5 | 7 | 5 | 8 | 9 | 9
nanogram x hour/milliliter (ng*hr/mL) | NA (NA) — At doses less than 1.6 mg, the AUC(0-∞) could not be reliably quantified. | NA (NA) — At doses less than 1.6 mg, the AUC(0-∞) could not be reliably quantified. | 60.6 (49) | 197 (38) | 393 (84) | 1680 (34) | 49.9 (41) | 102 (111) | 575 (62) | 38.6 (25) | 151 (54) | 1020 (50)

4. Secondary Outcome: Pharmacodynamic(PD) Biomarker: Plasma Minimum Amyloid-Beta Peptide (A-beta) 1-40 Concentration
Description: Plasma minimum A-beta 1-40 concentration or nadir concentration (Cnadir) is defined as the lowest concentration of plasma A-beta 1-40 following dose administration.
Time Frame: Part A Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 postdose; Part C Day 14: Predose 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 120, 168, and 216 postdose
Population: All participants in Part A, Periods 1-3 and Part C, Period 3, who received at least one dose of study drug and had evaluable PD data analyzed per protocol. Participants in Part B and D were not assessed per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter (pg/mL)
Groups:
- Part A Placebo: Single dose of placebo given PO in capsule form in Period 1-4.
- Part A 0.1mg LY3202626: Single dose 0.1mg LY3202626 given PO in Period 1 Cohort 1.
- Part A 1.6 mg LY3202626: Single dose of 1.6mg LY3202626 given PO in Period 2 Cohort 1.
- Part A 15mg LY3202626: Single dose of 15mg LY3202626 given PO in Period 3 and Period 4 Cohort 1.
- Part C Placebo: Multiple doses of placebo given PO once daily for 14 days.
- Part C 1mg LY3202626 QD: Multiple doses of 1mg LY3202626 in given PO once daily for 14 days.
Arm/Group | Part A Placebo | Part A 0.1mg LY3202626 | Part A 0.4mg LY3202626 | Part A 1.6 mg LY3202626 | Part A 5mg LY3202626 | Part A 15mg LY3202626 | Part A 45mg LY3202626 | Part C Placebo | Part C 1mg LY3202626 QD | Part C 6mg LY3202626 QD | Part C 26mg LY3202626 QD
Number analyzed (Participants) | 24 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 9 | 9 | 9
Picogram per milliliter (pg/mL) | 107 (35.1) | 58.1 (150) | 61.8 (25.6) | 33.4 (62.0) | 25.2 (16.8) | 17.0 (33.6) | 7.93 (42.0) | 84.6 (26.5) | 24.0 (33.1) | 5.80 (51.9) | 4.2 (0)

5. Secondary Outcome: PD Biomarker: Cerebral Spinal Fluid (CSF) Minimum Amyloid-beta Peptide (A-beta) 1-40 Concentration
Description: CSF minimum A-beta 1-40 concentration or nadir concentration (Cnadir) is defined as the lowest concentration of CSF A-beta 1-40 following dose administration.
Time Frame: Part B: -4, -2, Predose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 18, 20, 24, 28, 32, and 36 hours postdose
Population: All participants in Part B who received at least one dose of study drug and had evaluable CSF PD data analyzed per protocol. Participants in Part A, C and D were not assessed per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Part B Placebo: Single dose of placebo given PO in Period 1.
- Part B 1.6 mg LY3202626: Single dose of 1.6mg LY3202626 given PO in Period 1.
- Part B 6mg LY3202626: Single dose of 6mg LY3202626 given PO in Period 1.
Arm/Group | Part B Placebo | Part B 1.6 mg LY3202626 | Part B 6mg LY3202626 | Part B 26mg LY3202626
Number analyzed (Participants) | 3 | 5 | 5 | 5
pg/mL | 7980 (53.8) | 5700 (22.3) | 5770 (41.8) | 2980 (46.4)

6. Secondary Outcome: PK: CSF Concentration of LY3202626
Time Frame: Part C: Day 15 at 24 hours +/- 4 hours (hr) postdose
Population: All participants in Part C who received at least one dose of study drug and had evaluable CSF PK data per protocol. Participants in Part A, B and D were not assessed per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part C 1mg LY3202626: Multiple doses of 1mg LY3202626 given PO once daily for 14 days.
- Part C 6 mg LY3202626: Multiple doses of 6mg LY3202626 given PO once daily for 14 days.
- Part C 26mg LY3202626: Multiple doses of 26mg LY3202626 given PO once daily for 14 days.
Arm/Group | Part C 1mg LY3202626 | Part C 6 mg LY3202626 | Part C 26mg LY3202626
Number analyzed (Participants) | 9 | 9 | 9
ng/mL | 0.0648 (46.2) | 0.202 (48.9) | 1.26 (44.8)

7. Secondary Outcome: PD Biomarker: Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid-beta Peptide (A-beta) 1-40 Concentration
Description: CSF Aβ1-40 change from baseline at Day 15 endpoint, 24 hours postdose (+/- 4 hours) following multiple doses of LY3202626.
Time Frame: Parts C: Baseline, Day 15
Population: All participants in Part C who received at least one dose of study drug and had evaluable CSF PD data analyzed. Participants in Part A, B and D were not assessed per protocol.
Measure: Mean (Standard Deviation); unit: percent change in concentration
Groups:
- Part C 6mg LY3202626: Multiple doses of 6mg LY3202626 given PO once daily for 14 days.
Arm/Group | Part C Placebo | Part C 1mg LY3202626 | Part C 6mg LY3202626 | Part C 26mg LY3202626
Number analyzed (Participants) | 9 | 9 | 9 | 9
percent change in concentration | -21.3 (16.8) | -50.1 (8.56) | -75.7 (7.38) | -93.7 (2.39)

ADVERSE EVENTS:
Groups:
- Part A, B, and C Placebo: Single dose of placebo given PO in in capsule form, Part A and B. Multiple doses of placebo given PO in capsule form, Part C.
- Part A 0.1mg LY3202626: Single dose of 0.1mg LY3202626 given PO in in capsule form.
- Part A 0.4mg LY3202626: Single dose of 0.4mg LY3202626 given PO in in capsule form.
- Part A 0.4mg LY3202626 + 200mg Itraconazole: Single dose of 0.4mg LY3202626 +200mg Itraconazole given PO in in capsule form.
- Part C 1mg LY3202626 QD: Multiple daily dose of 1mg LY3202626 given PO in in capsule form.
- Part A and B 1.6mg LY3202626: Single dose of 1.6mg LY3202626 given PO in in capsule form..
- Part A 5mg LY3202626: Single dose of 5mg LY3202626 given PO in in capsule form.
- Part C and Part D 6mg LY3202626 QD: Multiple daily dose of 6mg LY3202626 given PO in capsule form.
- Part A and B 10mg LY3202626: Single dose of 10mg LY3202626 given PO in capsule form.
- Part A 15mg LY3202626: Single dose of 15mg LY3202626 given PO in capsule form.
- Part B and C 26mg LY3202626: Single dose of 26mg LY3202626 given PO in capsule form, Part B. Multiple daily dose of 26mg LY3202626 in in capsule form, Part C.
- Part A 45mg LY3202626: Single dose of 45mg LY3202626 given PO in in capsule form.
Arm/Group | Part A, B, and C Placebo | Part A 0.1mg LY3202626 | Part A 0.4mg LY3202626 | Part A 0.4mg LY3202626 + 200mg Itraconazole | Part C 1mg LY3202626 QD | Part A and B 1.6mg LY3202626 | Part A 5mg LY3202626 | Part C and Part D 6mg LY3202626 QD | Part A and B 10mg LY3202626 | Part A 15mg LY3202626 | Part B and C 26mg LY3202626 | Part A 45mg LY3202626
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/8 | 0/8 | 0/12 | 0/9 | 0/13 | 0/8 | 0/11 | 0/19 | 0/11 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 10/36 | 0/8 | 1/8 | 7/12 | 4/9 | 4/13 | 3/8 | 6/11 | 7/19 | 2/11 | 13/14 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, B, and C Placebo (N=36) | Part A 0.1mg LY3202626 (N=8) | Part A 0.4mg LY3202626 (N=8) | Part A 0.4mg LY3202626 + 200mg Itraconazole (N=12) | Part C 1mg LY3202626 QD (N=9) | Part A and B 1.6mg LY3202626 (N=13) | Part A 5mg LY3202626 (N=8) | Part C and Part D 6mg LY3202626 QD (N=11) | Part A and B 10mg LY3202626 (N=19) | Part A 15mg LY3202626 (N=11) | Part B and C 26mg LY3202626 (N=14) | Part A 45mg LY3202626 (N=8)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 9 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (8) | 0 (0) | 2 (2) | 5 (12) | 0 (0) | 5 (8) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days